CLINICAL TRIAL: NCT01723865
Title: Clinical Efficacy of a Specifically Dedicated Remote Monitoring System in the Management of Patients With Heart Failure and ICD&CRT-D.
Brief Title: Clinical Efficacy of Remote Monitoring in the Management of Heart Failure
Acronym: EFFECT
Status: Completed | Type: Observational
Sponsor: Effect Group, Italy (Network)
Responsible Party: Sponsor
Other Study IDs: Effect
Record Dates: First submitted 2012-10-23; First posted 2012-11-08 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Heart Failure
Keywords: Heart failure; Remote Monitoring; ICD; Follow-up
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conventional: Patients with heart failure having an ICD-CRT implanted, followed by conventional visits.
- Remote Monitoring: Patients with heart failure having an ICD-CRT implanted, followed by remote monitoring.

SUMMARY:
This is a clinical trial to evaluate the clinical benefit of remote monitoring in patients with heart failure having an ICD-CRT implanted.

Study purpose The purpose of this study is to test the hypothesis that the monitoring of specific clinical parameters, obtained by remote controls of ICD-CRT could improve clinical course of patients with heart failure.

Study design This is a prospective observational study, comparing clinical course of patients with heart failure having an ICD-CRT implanted, followed or not by remote monitoring. This study will include 870 subjects with ICD and CRT-D, and followed by a remote monitoring system (with or without weight and pressure external sensors) or followed by conventional ambulatory visits.

Primary endpoints The primary endpoint of this study is to document no superiority of unplanned hospital access for cardiac reasons (included access to the emergency units ) or death for cardiovascular causes in remote monitoring group (with or without weight and pressure external sensors) compared to conventional follow-up (usual care group).

DETAILED DESCRIPTION:
Aim of the study The purpose of this study is to evaluate the clinical benefit of a dedicated remote monitoring system (RPM) in the management of patients with heart failure and implanted with ICDs and CRT-D.

The clinical benefit will be assessed by:

* Increased cardiovascular events (death, myocardial infarction, hospitalization).
* Events arrhythmia: atrial fibrillation, sustained and nonsustained ventricular tachycardia or ventricular fibrillation.
* Autonomic profile, echocardiographic parameters, 6-minute walk test, quality of life questionnaire.

The primary endpoint of this study is to estimate the incidence (and its accuracy) of the first event of unplanned hospitalizations for cardiac reasons or death from cardiovascular causes in the group monitored using RPM (with or without external sensors) and in the group management via conventional follow-up (Usual Care).

ELIGIBILITY:
Inclusion Criteria:

* Subjects >18 years
* patients implanted or eligible for implant with ICD-CRT-D, accordingly with guidelines of the centers, for heart failure treatment and/or primary prevention of sudden death

Exclusion Criteria:

* Presence of clinically overt heart failure.
* Myocardial infarction within 2 months before enrolment.
* Significant concurrent illness or condition severely limiting life expectancy.
* Any surgical or medical condition which, at the discretion of the investigator, place the patient at higher risk from his/her participation in the study, or are likely to prevent the patient from complying with the requirements of the study or completing the trial period.
* History of drug or alcohol abuse within the last 2 years.
* Inability to communicate and comply with all study requirements including the unwillingness or inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both gender implanted or eligible for implant with ICD-CRT-D, for heart failure treatment and/or primary prevention of sudden death, followed or not by a remote monitoring system.
Sampling Method: Non-Probability Sample
Enrollment: 988 (Actual)
Dates: Start 2011-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
unplanned hospitalizations or death | 1 year
  unplanned hospitalization or for cardiac reasons or death for cardiovascular causes in the group monitored using RPM (with or without external sensors) and in the group management via conventional follow-up (Usual Care).

SECONDARY OUTCOMES:
All reasons hospitalizations | 1 year
Hospitalization for cardiac causes | 1 year
Myocardial infarction | 1 year
  Incidence of myocardial infarction
Ventricular tachycardia or fibrillation | 1 year
  Incidence of ventricular tachycardia or fibrillation
Atrial fibrillation | 1 year
  Incidence of atrial fibrillation episodes.
Heart transplantation | 1 year
  heart transplantation occurence
Cost for National Health System (NHS) | 1 year
  Estimate the total cost for the NHS for the management of heart failure patients implanted with ICD-CRT, monitored or not with a remote monitoring system.
Clinical benefit | 1 year
  Evaluate the clinical benefit by means of 6-minute walking test, use of medications and changes of echocardiographic parameters, between the patients followed by conventional visits and patients followed by remote controls (with or without external sensors).

OTHER OUTCOMES:
Autonomic activity | 1 year
  Indexes of autonomic activity such as th mean of standard deviations of RR intervals calculated on 5 minutes intervals (SDANN), activity log and "footprint", will be compared in patients followed by conventional visits of by remote controls.

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Buja, MD, Principal Investigator — University of Padova
Locations (16):
- Italy (16):
  - Ospedali riuniti di Ancona, Ancona
  - Azienda Ospededaliero Universitaria Policlinico, Bari
  - Ospedale di Venere, Bari
  - Ospedale S.Spirito, Casale Monferrato
  - Ferrari Hospital, Casarano
  - Presidio Ospedaliero Ferrari, Castrovillari
  - Policlinico V,Emanuele - Cardiologia Ferrarotto, Catania
  - Fondazione Istituto San Raffaele G.Giglio, Cefalù
  - Dep. of Cardiology, Civic Hospital, Cirié
  - Vito Fazzi Hospital, Lecce
  - Civic Hospital, Moncalieri
  - Ospedale dei Colli - Monaldi, Napoli
  - Clinica Mediterranea, Napoli
  - Ospedale dei Colli, Monaldi, Napoli
  - Dept. Cardiology, S. Cuore Hospital, Negrar
  - Dipartimento di Scienze Cardiologiche, Toraciche e Vascolari-Università di Padova, Padua

REFERENCES:
- [Derived] Capucci A, De Simone A, Luzi M, Calvi V, Stabile G, D'Onofrio A, Maffei S, Leoni L, Morani G, Sangiuolo R, Amellone C, Checchinato C, Ammendola E, Buja G. Economic impact of remote monitoring after implantable defibrillators implantation in heart failure patients: an analysis from the EFFECT study. Europace. 2017 Sep 1;19(9):1493-1499. doi: 10.1093/europace/eux017. PMID 28407139
- [Derived] De Simone A, Leoni L, Luzi M, Amellone C, Stabile G, La Rocca V, Capucci A, D'onofrio A, Ammendola E, Accardi F, Valsecchi S, Buja G. Remote monitoring improves outcome after ICD implantation: the clinical efficacy in the management of heart failure (EFFECT) study. Europace. 2015 Aug;17(8):1267-75. doi: 10.1093/europace/euu318. Epub 2015 Apr 4. PMID 25842271